CLINICAL TRIAL: NCT05362539
Title: Novel Urine-Based DNA Methylation Biomarkers for Urothelial Bladder Carcinoma Detection in Patients With Hematuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Lecturer of Urology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AS-4-2022
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer
Keywords: Urothelial bladder carcinoma; Bladder cancer; Hematuria; Biomarkers; DNA methylation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria | interventions — Cystoscopy; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hematuria patients (Experimental): Voided urine was collected from consecutive patients presented with hematuria at our institute for urine cytology and DNA hypermethylation assay of the assigned genes using methylation-specific Polymerase Chain Reaction (PCR). Further assessment by office cystoscopy and imaging with subsequent inpatient cystoscopic biopsy for positive findings, was done. The diagnostic characteristics of DNA hypermethylation and urine cytology were assessed based on its capability to predict UBC noninvasively
  Interventions: Procedure: Cystoscopy; Diagnostic Test: Computed tomography; Genetic: DNA hypermethylation assay; Diagnostic Test: Urine cytology

INTERVENTIONS:
Procedure: Cystoscopy — diagnostic cystoscopy for detection of any bladder lesions
Diagnostic Test: Computed tomography — Computed tomography for patients to exclude bladder lesions
Genetic: DNA hypermethylation assay — DNA hypermethylation assay of six genes (GATA4, P16, P14, APC, CDH1 and CD99)
Diagnostic Test: Urine cytology — voided urine cytology for all patients

SUMMARY:
The current study aimed to assess the diagnostic performance of novel urine-based DNA hypermethylation of six genes (GATA4, P16, P14, APC, CDH1 and CD99) for UBC detection in patients with hematuria.

DETAILED DESCRIPTION:
According to GLOBOCAN data, bladder cancer (BC) is considered a major health problem that represents 3% of all cancer diagnoses. Urothelial bladder carcinoma (UBC) accounts for the vast majority (>90%) of BC cases with predominance of non-muscle invasive disease (Ta, Tis or T1) in 75% of patients while others show muscle invasion (T2-4).

In refereed population, UBC is usually diagnosed as a result of work-up for hematuria at a rate of 2-5% following an evaluation of asymptomatic microscopic hematuria, and, up to 5-15% of patients with macroscopic hematuria. Therefore, a timely prompt evaluation of hematuria can give to earlier diagnosis and better survival of UBC.

Currently, cystoscopy /cross sectional imaging are the gold standard tools for UBC diagnosis in patients with hematuria. Unfortunately, these costly, invasive and painful diagnostics could miss early, small/flat bladder lesions. Urine cytology has been proposed as a non-invasive alternative test with high specificity, however, it lacks sensitivity for diagnosis of low grade (LG) tumors.

Over the last decades, multiple researches have output different markers for UBC diagnosis. Based on their target of assessment, these markers include screening for soluble antigens (BTA-Stat, NMP-22, surviving, etc.), cell surface antigens (Cytokeratins and UroVysion), genomic markers (Cxbladder and Xpert) and urinary metabolomics (CRAT and SLC25A20). However, most of these markers are limited by unsatisfying diagnostic performance, high cost or lack of validation.

Several preliminary studies have shown that DNA methylation, a critical step in transcription regulation, is chemically stable and can be precisely quantified, making it an attractive marker for UBC detection. Both local and global DNA hypermethylation in BC specimens are usually associated with inactivation of tumor suppressor genes. These methylations changes could be effectively identified in urine sediments as well as tumor tissues.

In the current literature, multiple studies investigated the performance of DNA hypermethylation of either individual or panel genes with reported sensitivity (SN) and specificity (SP) values that range from 40-95 % and 10-100 %, respectively. Most of these studies were limited by tumor characteristics heterogeneity (majority were ≥T2 and high grade (HG) disease; which did not reflect the daily practice, inclusion of different BC histological variants), lack of external validation and small sample size.

The aim of our study is to assess the diagnostic performance of novel urine-based DNA methylation six genes (GATA4, P16, P14, APC, CDH1 and CD99) for UBC detection in patients with hematuria. Moreover, we investigated the methylation pattern of these genes in different stages and grades of UBC.

ELIGIBILITY:
Inclusion Criteria:

* patients with hematuria (macroscopic or microscopic)

Exclusion Criteria:

* history of Bladder Cancer
* history of pelvic irradiation,
* bleeding diathesis or receiving anticoagulants
* patients with upper urinary tract neoplasm or urolithiasis

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of hypermethylation of six genes (GATA4, P16, P14, APC, CDH1 and CD99) in patients with urothelial bladder carcinoma | 4 weeks
  Rate of hypermethylation of six genes (GATA4, P16, P14, APC, CDH1 and CD99) in patients with urothelial bladder carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No